CLINICAL TRIAL: NCT03826238
Title: Alcohol Related Brain Damage: Exploring Virtual Reality Based Cognitive Function Assessment and EEG Biomarkers. A Pilot Study
Brief Title: VR Assessment for Alcohol Related Brain Damage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Institute for Bioengineering of Catalonia (Other)
Responsible Party: Principal Investigator, Paul Verschure, Principal Investigator, Universitat Pompeu Fabra
Other Study IDs: REHABOH-VG
Record Dates: First submitted 2018-11-08; First posted 2019-02-01 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Alcohol-Related Disorders
Keywords: alcohol-related brain damage; depression; attention; eeg
MeSH Terms: conditions — Alcohol-Related Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ARBD and depression: 10 patients with ARBD and at least moderate depressive symptoms (MoCA < 26, Hamilton Depression Rating Scale ≥ 17). Intervention: The Validation Gate task, a visual attention task where the subject must detect discontinuities in the moving trajectory of circles on the screen while EEG is recorded.
  Interventions: Diagnostic Test: Validation Gate task
- ARBD and no depression: 10 patients with ARBD and no clinically relevant depressive symptoms (MoCA < 26, Hamilton Depression Rating Scale < 17). Intervention: The Validation Gate task, a visual attention task where the subject must detect discontinuities in the moving trajectory of circles on the screen while EEG is recorded.
  Interventions: Diagnostic Test: Validation Gate task
- Healthy: 10 healthy controls (no ARDB, no depression, no cognitive deficit). Intervention: The Validation Gate task, a visual attention task where the subject must detect discontinuities in the moving trajectory of circles on the screen while EEG is recorded.
  Interventions: Diagnostic Test: Validation Gate task

INTERVENTIONS:
Diagnostic Test: Validation Gate task — The task is to observe several moving unfilled white circles on a dark background. The circles move in straight paths. Every so often, a randomly selected circle will displace to a point inconsistent with its trajectory, which will look like a "jump". The subjects' task is to press the space bar every time they detect a displacement (e.g. jump). A session consists of 30 minutes, it starts with 2 training blocks which are followed by 2 no-cognitive load blocks and 6 blocks with increasing cognitive load conditions. During the assessment the eye movement as well as the key presses are registered in order to calculate early and late saccades as well as conscious reporting. Resting-state EEG will also be recorded and compared to the ones of age-matched healthy controls. Task-dependent EEG data will be recorded during the Validation Gate task.

SUMMARY:
Pilot study where 10 alcohol-related brain damage (ARBD) patients will undergo a 30-minutes-long cognitive assessment session using the Validation Gate task to evaluate usability of this tool in Alcohol Use Disorder patients. Resting-state EEG of ARBD patients will also be recorded and compared to the ones of age-matched healthy people in order to preliminary explore the existence of possible EEG biomarkers of ARBD.

DETAILED DESCRIPTION:
Much of the burden of disease related to harmful alcohol use is due to the persistent effects of alcohol on central nervous system. The concept of alcohol-related brain damage (ARBD) is important in the Addiction Psychiatry field. ARBD is a spectrum of disorders. Besides most severe forms, 50-70% of patients with alcohol use disorder suffer some kind of cognitive impairment, being mild to moderate cognitive impairment the most frequent disorders, and often the most difficult to detect. In alcoholic patients, greater cognitive impairment has been associated with less treatment compliance and fewer days of abstinence. Considering its impact, cognitive screening should be enhanced.

Recently, standard assessments have been augmented with new interactive technology. The work group of the Laboratory of Synthetic, Perceptive, Emotive and Cognitive Systems (SPECS), part of Institute for Bioengineering of Catalonia (IBEC), developed a virtual assessment of cognitive function, called the Validation Gate task, which evaluates sustained attention, working memory and executive functioning. This tool has been used so far in chronic stroke patients, showing that, in this group, depression symptoms affect performance in this task.

Similarly to chronic stroke patients, a diffuse harm of several cognitive domains in ARBD is observed. In the addiction psychiatry field, the gold standard to evaluate changes in cognitive function are still thorough neuropsychological test batteries. But performing thorough neuropsychological evaluations on all patients in daily clinical practice is highly resource consuming (need of expert neuropsychologists, time consuming). These last years scientific community has also been trying to find biomarkers of ARBD in electrophysiological tests, with no conclusive results.

In this pilot study a small number of ARBD patients and healthy people will undergo a single 30-minutes-long cognitive assessment session using the Validation Gate task to evaluate usability of this tool in Alcohol Use Disorder patients. Resting-state EEG of ARBD patients will also be recorded and compared to the ones of age-matched healthy controls in order to preliminary explore the existence of possible EEG biomarkers of ARBD.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Use Disorder (DSM 5) as main substance
* Positive screening for alcohol related cognitive impairment (Montreal Cognitive Assessment, MoCA < 26)
* abstinent during 15 to 90 days according to self-reports
* no severe upper limb motor disability.
* Older than 18 years old.
* abìlity to talk, understand and write in Catalan, Spanish or English.
* sign informed consent

Exclusion Criteria:

* severe cognitive incapacity that prohibits the execution of the assessment
* severe impairments like spasticity, communication disabilities (aphasia or apraxia) and perceptual or physical impairments that would interfere with the correct execution or understanding of the assessment
* history of other serious mental-health problems in acute or subacute phase
* comorbidity with severe neurological illness
* regular use of other substances (except nicotine)
* active intake of benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ARBD (Groups A and B) will be consecutively recruited from the Addiction outpatient and Day Hospital Unit of Addiction Unit at the Department of Psychiatry at Hospital Clínic in Barcelona.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Virtual assessment (Validation Gate task) | 30 minutes
  The Validation Gate task, a visual attention task where the patient must detect discontinuities in the moving trajectory of circles on the screen. In this task the following variables will be registered: fast and slow eye saccades as well as conscious detections.
Montreal Cognitive Assessment (MoCA) | 20 minutes
  MoCA test is a screening test for cognitive impairment that explores 8 domains: visuospatial/executive ability, naming, memory, attention, language, abstraction, delayed recall, and orientation.
Hamilton Depression Rating Scale | 10 minutes
  Evaluation tool of depression. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. The summed score indicates severity (0-7 no depression, > 23 very severe depression)

SECONDARY OUTCOMES:
Resting State and task-dependent EEG | 40 minutes
  6 minutes of EEG data during resting state and 30 minutes of EEG during the Validation Gate taks, will be acquired through the wireless sensor system ENOBIO32 of Starlab. From these recordings the mean spectral energy in the common frequency bands will be obtained as variables to identify signatures of TCD and the theta activity in the different groups.
The alcohol, smoking and substance involvement screening test (ASSIST) | 10 minutes
  The ASSIST scale is used to detect substance use and classify risk and severity for each substance. Each question (8 questions) on the ASSIST has a set of responses to choose from, and each response has a numerical score (for instance they can range from 0 for "never" to up to 8 for "daily"). The interviewer simply circles the numerical score that corresponds to the patient's response for each question/substance. At the end of the interview the scores for each substance are added together to produce an ASSIST score for that substance. Low numbers mean low risk, high numbers mean high risk. We are testing only for "Alcohol-Risk", which can have a risk-score from 0 to 31.
Alcohol Use Disorders Identification Test (AUDIT) | 10 minutes
  Assessment of alcohol use

CONTACTS AND LOCATIONS:
Locations (1):
- Addictions Unit. Psychiatry and Psychology Service. Institut Clínic de Neurociències (ICN). Hospital Clínic de Barcelona. IDIBAPS, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
For the moment IDP is shared between the involved investigators at Hospital Clínic de Barcelona and IBEC.